CLINICAL TRIAL: NCT01244555
Title: Muscle Treatment for Management of Pain & Disability in Tension-type Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0085; 1R21AT004469-01A2 (NIH)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Tension-type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — High-Energy Shock Waves; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Massage treatment (Experimental)
  Interventions: Other: massage
- Ultrasound (Experimental)
  Interventions: Other: ultrasound
- Wait-list (No Intervention)

INTERVENTIONS:
Other: ultrasound — Twice weekly ultrasound sessions for 6 weeks
  Arms: Ultrasound
Other: massage — Twice weekly massage sessions for 6 weeks
  Other Names: myofsacial trigger point therapy
  Arms: Massage treatment

SUMMARY:
The purpose of this study is to determine the effectiveness of treatments (massage therapy or ultrasound) directed at skeletal muscle for alleviating pain associated wtih tension headache.

DETAILED DESCRIPTION:
Chronic or episodic forms of tension-type headache affect a high percentage of the population. Pain from tension-type headache (TTH) not only impacts personal well-being, but also poses a significant socioeconomic burden in terms of workdays lost and decreased worker productivity. Although TTH is the most prevalent of the headache disorders, there is a distinct lack of research with regards to specific treatments for this ailment in comparison to all other headache classifications, such as migraine. A muscular involvement is associated with TTH and is reported in the research literature as elevation in skeletal muscle tenderness, increased presence of active myofascial trigger point's, and physical abnormalities in cervical and cranial muscles. Thus, a treatment approach that addresses the skeletal musculature could be an important component in the management of TTH. The purpose of this randomized trial is to determine the effectiveness of two muscle oriented treatments on reducing pain and disability associated with TTH: massage therapy and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more tension-type headache episodes per week
* Headache episodes of 2 hours or longer
* Experiencing tension-type headache for 6 months or longer

Exclusion Criteria:

* Migraine >1/month
* Presence of alternate forms of headache (e.g. cluster headache, medication-induced headache, headache caused by injury)
* The diagnosis of fibromyalgia, major depression, other neurological or cardiovascular disease
* Pregnancy
* Prior massage or ultrasound treatment for headaches

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Headache frequency | Measure is assessed daily for 14 weeks

SECONDARY OUTCOMES:
Headache Disability Index | Assessed at 4 time points over 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moraska, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States